CLINICAL TRIAL: NCT01223014
Title: An Open Label, Single Dose, Phase I Study to Evaluate the Excretion of Radioactivity, the Metabolic Profile, Pharmacokinetics, Safety and Tolerability Following Single Oral Administration of [14C]AZD2423 to Healthy Male Volunteers
Brief Title: Study Evaluating Absorption, Distribution, Metabolism and Excretion (ADME) of Single Dose [14C] AZD2423 in Volunteers
Acronym: ADME
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Marketing Company Medical Director, AstraZeneca
Other Study IDs: D2600C00008
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Neuroscience
Keywords: Radioactive; ADME; Neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pharmacogenetic samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Single cohort of 6 subjects
  Interventions: Drug: AZD2423

INTERVENTIONS:
Drug: AZD2423 — AZD2423

SUMMARY:
Phase I study to evaluate the excretion of radioactivity, the metabolic profile, pharmacokinetics, safety and tolerability following a single oral administration of [14C]AZD2423 in healthy male volunteers aged 50 to 65 years (inclusive).The purpose of this study is to investigate how and how quickly AZD 2423 or its break down products are excreted by analysing blood, faeces and urine samples collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥18 and ≤30 kg/m2 and weight of ≥50 kg and ≤100 kg
* Regular daily bowel movements (ie, production of at least 1 stool per day)
* Provision of signed and dated, written informed consent prior to any study specific procedures

Exclusion Criteria:

* Healthy volunteers exposed to radiation levels above background (eg, through X ray examination) of >5 mSv in the last year, >10 mSv over the last 5 years or a cumulative total of >1 mSv per year of life
* Participation in any prior radiolabelled study within 12 months of the screening visit (Visit 1)
* History of alcohol abuse or excessive intake of alcohol defined as regular intake of more than 15 units of alcohol a week. (unit = 1 glass of wine (125 mL) = 1 measure of spirits = ½ pint of beer)

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic/community sample
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 1
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 2
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 3
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 4
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 5
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 6
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 7
Percentage of radioactive dose recovered in urine and faeces and total percentage | During residential period on Day 8
Concentration of total radioactivity in blood and plasma | During residential period on Day 1
Concentration of total radioactivity in blood and plasma | During residential period on Day 2
Concentration of total radioactivity in blood and plasma | During residential period on Day 3
Concentration of total radioactivity in blood and plasma | During residential period on Day 4
Concentration of total radioactivity in blood and plasma | During residential period on Day 5
Concentration of total radioactivity in blood and plasma | During residential period on Day 6
Concentration of total radioactivity in blood and plasma | During residential period on Day 7
Concentration of total radioactivity in blood and plasma | During residential period on Day 8

SECONDARY OUTCOMES:
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing adverse events | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing concomitant medications | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing clinical chemistry | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing haematology | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing urinalysis | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing vital signs | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing body weight | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by assessing electrocardiogram | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of AZD2423 following administration of a single oral dose of [C14] AZD2423 solution by physical examination | Range of Day -1 until follow up visit (Visit 3)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Lilja, Study Director — AstraZeneca; Marianne Kasti, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London, United Kingdom